CLINICAL TRIAL: NCT06877975
Title: Validation and Testing of a Novel CGM-CKM Device in Healthy Volunteers
Brief Title: Validation and Testing of a Novel Continuous Glucose and Continuous Ketone Monitoring Device in Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Mahla Poudineh, Assistant Professor, University of Waterloo
Other Study IDs: 46561; 2-SRA-2022-1167-M-B (Other Grant/Funding Number: Breakthrough T1D)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for glucose and ketone measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals

SUMMARY:
Diabetic ketoacidosis (DKA) is a severe complication of type 1 diabetes (T1D) that can have life-threatening consequences. It occurs when there is a high level of glucose in the blood and the body produces excessive amounts of ketone bodies. To manage this condition, individuals with T1D need to constantly monitor their levels of ketone bodies and glucose. While continuous glucose monitoring (CGM) devices have made significant advancements in providing non-invasive or minimally invasive glucose measurements, there has been little progress in developing methods for continuous monitoring of ketone bodies (CKM). Currently, the commonly used approaches involve self monitoring with commercially available blood or urine strips. However, these tools have limited adoption, provide only single time point measurements, and can be costly for some patients.

In our project, which is funded by Breakthrough T1D (2-SRA-2022-1167-M-B), we address this challenge by utilizing a minimally invasive biosensor based on hydrogel microneedle (HMN). This biosensor enables simultaneous and continuous measurement of the primary biomarker for ketone formation, 3-β hydroxybutyrate (β-HB), as well as glucose levels. By doing so, we intend to reduce the risk of diabetic ketoacidosis in patients with T1D. We plan to test the developed CGM-CKM device on human subjects, including both healthy volunteers (HV) and patients with T1D. The HV testing will take place at the laboratory of Dr. Poudineh and Dr. Devries-Aboud in Waterloo, while the validation involving patients with T1D will be conducted in collaboration with Dr. Lal at Stanford.

ELIGIBILITY:
The age range for the healthy volunteers (HVs) will be between 18 and 45 years old and with no family history of Diabetes (T1D or T2D, specifically biological parents and siblings).

Exclusion criteria included: (i) currently taking any medications (except for birth control for females); (ii) following a low-carbohydrate diet or consuming nutritional ketone supplements; (iii) considered competitive athlete engaged in competition or intensive training, (iv) have been diagnosed with Diabetes (T1D or T2D), hypertension, cardiovascular disease, kidney disease, and thyroid disorder. (v) Having an allergy to any of the ingredients in the products used in the study, which will be explained to you in detail.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers (HVs) will be between 18 and 45 years old and with no family history of Diabetes (T1D or T2D, specifically biological parents and siblings).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of the sensor measurement with blood-based measurement | 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Sensor measurements and blood glucose and ketone levels will be shared via publications.

REFERENCES:
- [Result] GhavamiNejad P, GhavamiNejad A, Zheng H, Dhingra K, Samarikhalaj M, Poudineh M. A Conductive Hydrogel Microneedle-Based Assay Integrating PEDOT:PSS and Ag-Pt Nanoparticles for Real-Time, Enzyme-Less, and Electrochemical Sensing of Glucose. Adv Healthc Mater. 2023 Jan;12(1):e2202362. doi: 10.1002/adhm.202202362. Epub 2022 Oct 13. PMID 36183355
- [Result] Ausri IR, Sadeghzadeh S, Biswas S, Zheng H, GhavamiNejad P, Huynh MDT, Keyvani F, Shirzadi E, Rahman FA, Quadrilatero J, GhavamiNejad A, Poudineh M. Multifunctional Dopamine-Based Hydrogel Microneedle Electrode for Continuous Ketone Sensing. Adv Mater. 2024 Aug;36(32):e2402009. doi: 10.1002/adma.202402009. Epub 2024 Jun 16. PMID 38847967